CLINICAL TRIAL: NCT01486355
Title: A Randomised Trial of an Additional Measles Vaccine at 4 Months of Age to Reduce Child Mortality and to Explore the Role of Maternal Measles Antibodies for the Beneficial Non-specific Effects of Measles Vaccine
Brief Title: Additional Measles Vaccine at 4 Months of Age
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bandim Health Project (Other)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: MVurban
Record Dates: First submitted 2011-08-03; First posted 2011-12-06 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Measles Infection
Keywords: Mortality; Morbidity; Hospitalisations/consultations; Growth; Measles infection
MeSH Terms: interventions — Measles Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early measles vaccine (Experimental): Receives an early measles vaccine in addition to the standard measles vaccine at 9 months of age
  Interventions: Biological: Measles vaccine
- No early measles vaccine (No Intervention): Receives only the standard measles vaccine at 9 months of age

INTERVENTIONS:
Biological: Measles vaccine — Edmonston-Zagreb measles vaccine
  Arms: Early measles vaccine

SUMMARY:
Overall objective: To conduct a randomised controlled trial (RCT) to examine whether an early two-dose measles vaccination (MV) strategy at 4 and 9 months will reduce child mortality compared with the WHO strategy of one dose of MV at 9 months.

Specific hypotheses Hypothesis I) Two doses of MV at 4 and 9 months compared with the standard dose of MV at 9 months will reduce mortality by 30% between 4 months and 5 years of age1. As in a previous trial it is expected that the beneficial effect is strongest for girls.

Hypothesis II) Children receiving MV at 4 months in the presence of maternal measles antibodies (MatAb) will have 35% lower mortality between 4 months and 5 years of age than children receiving MV at 4 months with no detectable MatAb.

Implications: These hypotheses are based on a previous RCT showing strong beneficial effects of providing an early measles vaccine, in particular among children with MatAb.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 7 months who received the third dose of pentavalent vaccine at least 4 weeks earlier

Exclusion Criteria:

* Malformations
* Severely ill
* Severely malnourished

Ages: 4 Months to 7 Months | Sex: All
Age Groups: Child
Dates: Start 2011-08; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Mortality
  Differences in mortality rates between the intervention and control groups

SECONDARY OUTCOMES:
Morbidity
  Symptoms of infection
Hospitalisations/consultations
  Visits to health center for consultation due to illness, hospitalisation
Growth
  Weight, length, arm circumference
Measles infection
  Measles infection assessed by medical doctor and/or verified by blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Bissau, Bissau Region, Guinea-Bissau

REFERENCES:
- [Background] Aaby P, Martins CL, Garly ML, Bale C, Andersen A, Rodrigues A, Ravn H, Lisse IM, Benn CS, Whittle HC. Non-specific effects of standard measles vaccine at 4.5 and 9 months of age on childhood mortality: randomised controlled trial. BMJ. 2010 Nov 30;341:c6495. doi: 10.1136/bmj.c6495. PMID 21118875
- [Derived] Nielsen S, Fisker AB, da Silva I, Byberg S, Biering-Sorensen S, Bale C, Barbosa A, Bjerregaard-Andersen M, Hansen NS, Do VA, Baek O, Rasmussen SM, Damkjaer L, Hvidt S, Baltzersen O, Rodrigues A, Martins C, Jensen KJ, Whittle HC, Smits G, van der Klis F, Aaby P, Benn CS. Effect of early two-dose measles vaccination on childhood mortality and modification by maternal measles antibody in Guinea-Bissau, West Africa: A single-centre open-label randomised controlled trial. EClinicalMedicine. 2022 May 27;49:101467. doi: 10.1016/j.eclinm.2022.101467. eCollection 2022 Jul. PMID 35747181
- [Derived] Hansen NS, Byberg S, Hervig Jacobsen L, Bjerregaard-Andersen M, Jensen AKG, Martins C, Aaby P, Skov Jensen J, Benn CS, Whittle H. Effect of early measles vaccine on pneumococcal colonization: A randomized trial from Guinea-Bissau. PLoS One. 2017 May 17;12(5):e0177547. doi: 10.1371/journal.pone.0177547. eCollection 2017. PMID 28545041
- [Derived] Christensen LD, Eriksen HB, Biering-Sorensen S, Bale C, Do VA, Andersen A, Martins CL, Sodemann M, Aaby P, Benn CS. The effect of early measles vaccination on thymic size. A randomized study from Guinea-Bissau. Vaccine. 2014 Mar 26;32(15):1641-4. doi: 10.1016/j.vaccine.2014.01.034. Epub 2014 Feb 9. PMID 24522160
- See also: Related Info — http://www.bandim.org